CLINICAL TRIAL: NCT02803827
Title: Optimizing the Management of Pediatric Acute Diarrhoeal Disease in Botswana
Brief Title: Optimizing the Management of Acute Diarrhoeal Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hamilton Health Sciences Corporation (Other)
Collaborators: Grand Challenges Canada (Other); BioMérieux (Industry); BioGaia AB (Industry); Copan Italia S.A. (Unknown); Botswana-UPenn Partnership (Other); University of British Columbia (Other)
Responsible Party: Principal Investigator, Jeffrey Pernica, Head, Division of Infectious Diseases, McMaster University
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GCC 0768-05
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2019-02-26 (Actual); Status verified 2019-02

CONDITIONS: Acute Gastroenteritis
Keywords: diarrhoea; gastroenteritis; rapid diagnostics; probiotics
MeSH Terms: conditions — Diarrhea; Gastroenteritis | interventions — Rapid Diagnostic Tests; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Rapid diagnostics and probiotic (Experimental): Participants randomized to this arm will have rapid enteric diagnostics performed on the day of enrolment. Those found to have a treatable pathogen will be prescribed antimicrobials that day. Participants will also be given Lactobacillus reuteri DSM 17938 5 x 10e8 cfu/mL x 60 days.
  Interventions: Other: Rapid diagnostics; Biological: Probiotic
- Rapid diagnostics and placebo (Other): Participants randomized to this arm will have rapid enteric diagnostics performed on the day of enrolment. Those found to have a treatable pathogen will be prescribed antimicrobials that day. Participants will also be given placebo x 60 days.
  Interventions: Other: Rapid diagnostics; Other: Placebo
- No rapid diagnostics and probiotic (Other): Participants randomized to this arm will have stool specimens processed after the conclusion of the study. Participants will also be given Lactobacillus reuteri DSM 17938 5 x 10e8 cfu/mL x 60 days.
  Interventions: Biological: Probiotic
- No rapid diagnostics and placebo (Placebo Comparator): Participants randomized to this arm will have stool specimens processed after the conclusion of the study. Participants will also be given placebo x 60 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Rapid diagnostics — Participants will have enteric specimens obtained using a flocked rectal swab, which will be transported in 2 mL Cary Blair medium. These will be tested using the BioMerieux BioFire FilmArray GI panel.
  Arms: Rapid diagnostics and placebo; Rapid diagnostics and probiotic
Biological: Probiotic — The probiotic given will be Lactobacillus reuteri DSM 17938, 5x10e8 cfu/mL x 60 days, suspended in vegetable oil.
  Arms: No rapid diagnostics and probiotic; Rapid diagnostics and probiotic
Other: Placebo — The placebo will be the vegetable oil vehicle and look identical to the probiotic.
  Arms: No rapid diagnostics and placebo; Rapid diagnostics and placebo

SUMMARY:
Many children admitted to hospital in Botswana without bloody diarrhoea are presumed to have viral gastroenteritis and so not treated with antibiotics - but they may indeed have a treatable cause for their illness. The investigators will conduct a randomized trial to see if rapid testing using novel methods to identify potentially treatable causes of diarrhoea leads to improved outcomes. The investigators will also be randomizing children to Lactobacillus reuteri DSM (daughter strain) 17938 therapy versus placebo (the standard of care) to see if this treatment decreases the duration of diarrhoea. The proposed study is a large multi-centre trial following the previous pilot trial.

ELIGIBILITY:
Inclusion Criteria:

* acute diarrhoeal illness (>= 3 stools in 24 hour period)

Exclusion Criteria:

* diarrhoeal illness >=14 days
* bloody stool
* known inflammatory bowel disease, cystic fibrosis, or malignancy
* live in a household with someone else documented to have a bacterial or parasitic enteric infection of defined aetiology
* live outside catchment areas
* no permanent address
* no access to mobile phone
* previous participation in this study
* nosocomial diarrhoea

Ages: 2 Months to 60 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 276 (Actual)
Dates: Start 2016-06; Primary Completion 2019-01 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
Height z-score (HAZ) adjusted for baseline HAZ | 60 days post-enrollment

SECONDARY OUTCOMES:
Mortality | 60 days post-enrollment
Weight z-score (WAZ) adjusted for baseline WAZ | 60 days post-enrollment
Environmental enteropathy score (EES) | 60 days
  composite of stool neopterin, myeloperoxidase, and alpha-1-antitrypsin
Diarrhoea recurrence | 60 days after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Pernica, MD, Principal Investigator — McMaster University
Locations (4):
- Botswana (4):
  - Princess Marina Hospital, Gaborone
  - Deborah Retief Hospital, Mochudi
  - Scottish Livingstone Hospital, Molepolole
  - Bamalete Lutheran Hospital, Ramotswa

REFERENCES:
- [Derived] Guitor AK, Katyukhina A, Mokomane M, Lechiile K, Goldfarb DM, Wright GD, McArthur AG, Pernica JM. Minimal Impact on the Resistome of Children in Botswana After Azithromycin Treatment for Acute Severe Diarrheal Disease. J Infect Dis. 2024 Jul 25;230(1):239-249. doi: 10.1093/infdis/jiae049. PMID 39052715
- [Derived] Pernica JM, Arscott-Mills T, Steenhoff AP, Mokomane M, Moorad B, Bapabi M, Lechiile K, Mangwegape O, Batisani B, Mawoko N, Muthoga C, Vanniyasingam T, Ewusie J, Lowe A, Bonsu JM, Gezmu AM, Smieja M, Mazhani L, Stordal K, Thabane L, Kelly MS, Goldfarb DM. Optimising the management of childhood acute diarrhoeal disease using a rapid test-and- treat strategy and/or Lactobacillus reuteri DSM 17938: a multicentre, randomised, controlled, factorial trial in Botswana. BMJ Glob Health. 2022 Apr;7(4):e007826. doi: 10.1136/bmjgh-2021-007826. PMID 35418412